CLINICAL TRIAL: NCT02618499
Title: Is Placental Transfusion Influenced by the Early Administration of Oxytocin?
Brief Title: Delayed Cord Clamping and Use of Oxytocin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility suggested by DSMC
Sponsor: Fundacion para la Salud Materno Infantil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Funda05
Record Dates: First submitted 2015-11-10; First posted 2015-12-01 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Placental Transfusion
Keywords: birth; oxytocin; placental transfusion; umbilical cord clamping
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxytocin inmediately at birth (Active Comparator): Intervention: Timing of administration of postpartum Oxytocin. 10 international Units (IU) immediately at birth will be given intravenously (IV) to the mother.
  Interventions: Drug: Timing of administration of post partum Oxytocin
- oxytocin at 3 minutes (Experimental): Intervention: Timing of administration of postpartum Oxytocin. 10 IU IV at 3 minutes immediately after the cord is clamped
  Interventions: Drug: Timing of administration of post partum Oxytocin

INTERVENTIONS:
Drug: Timing of administration of post partum Oxytocin — 10 IU of oxytocin given IV at different times after birth
  Other Names: syntosinon

SUMMARY:
The purpose of this study is to determine if oxytocin administration immediately after delivery of the infant modifies the volume of placental transfusion in healthy term infants.

DETAILED DESCRIPTION:
Randomized controlled trial with 2 arms to test the influence of oxytocin in placental transfusion.

Placental transfusion: the amount of blood that passes to the baby from the time of birth until the cord is clamped.

The difference in weight between a measurement at birth and a second one after clamping the cord at 3 minutes will be considered as proxy for placental transfusion.

In one arm the oxytocin will be used immediately after birth and the cord clamped at 3 minutes In the other arm the oxytocin will be administered at 3 minutes of birth after the cord is clamped.

ELIGIBILITY:
Inclusion Criteria:

* Healthy single Term pregnancies.
* Vaginal delivery.
* Informed consent obtained.
* Presence of an investigator

Exclusion Criteria:

* Placenta previa.
* Previous history of Postpartum hemorrhage
* Intrauterine growth restriction .
* Major congenital malformations.
* Eclampsia
* Extraction of blood sample for bank of umbilical cord stem cells.

Elimination criteria:

* Need for immediate assistance of the newborn
* Birth weight less than 2500 g
* Nuchal cord wrapped too tight
* Surgically finished delivery
* Short umbilical cord which might prevent placing the infant on the scale
* Technical difficulties to obtain the weight

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
placental transfusion | between birth and 3 minutes of life
  Difference in body weight between birth and 3 minutes of life

SECONDARY OUTCOMES:
bilirubin | at 36/48 hours
  Bilirubin level
Hematocrit | at 36/48 hours
  Hematocrit levels
Maternal blood loss | after birth for 30 minutes
  measure of the blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Vain, MD, Study Director — Fundasamin; Daniela S Satragno, MD, Principal Investigator — Fundasamin
Locations (1):
- Instituto de Ginecologia y Maternidad Nuestra Señora de la Merced, San Miguel de Tucumán, Tucumán Province, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonald SJ, Middleton P, Dowswell T, Morris PS. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2013 Jul 11;2013(7):CD004074. doi: 10.1002/14651858.CD004074.pub3. PMID 23843134
- [Background] Vain NE, Satragno DS, Gorenstein AN, Gordillo JE, Berazategui JP, Alda MG, Prudent LM. Effect of gravity on volume of placental transfusion: a multicentre, randomised, non-inferiority trial. Lancet. 2014 Jul 19;384(9939):235-40. doi: 10.1016/S0140-6736(14)60197-5. Epub 2014 Apr 17. PMID 24746755
- [Background] Westhoff G, Cotter AM, Tolosa JE. Prophylactic oxytocin for the third stage of labour to prevent postpartum haemorrhage. Cochrane Database Syst Rev. 2013 Oct 30;(10):CD001808. doi: 10.1002/14651858.CD001808.pub2. PMID 24173606
- [Background] Lalonde A; International Federation of Gynecology and Obstetrics. Prevention and treatment of postpartum hemorrhage in low-resource settings. Int J Gynaecol Obstet. 2012 May;117(2):108-18. doi: 10.1016/j.ijgo.2012.03.001. No abstract available. PMID 22502595
- [Background] Soltani H, Hutchon DR, Poulose TA. Timing of prophylactic uterotonics for the third stage of labour after vaginal birth. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD006173. doi: 10.1002/14651858.CD006173.pub2. PMID 20687079
- [Background] Begley CM, Gyte GM, Devane D, McGuire W, Weeks A. Active versus expectant management for women in the third stage of labour. Cochrane Database Syst Rev. 2015 Mar 2;(3):CD007412. doi: 10.1002/14651858.CD007412.pub4. PMID 25730178
- [Background] Yao AC, Hirvensalo M, Lind J. Placental transfusion-rate and uterine contraction. Lancet. 1968 Feb 24;1(7539):380-3. doi: 10.1016/s0140-6736(68)91352-4. No abstract available. PMID 4169972
- [Background] Farrar D, Airey R, Law GR, Tuffnell D, Cattle B, Duley L. Measuring placental transfusion for term births: weighing babies with cord intact. BJOG. 2011 Jan;118(1):70-5. doi: 10.1111/j.1471-0528.2010.02781.x. Epub 2010 Nov 18. PMID 21083868
- [Background] Trudnowski RJ, Rico RC. Specific gravity of blood and plasma at 4 and 37 degrees C. Clin Chem. 1974 May;20(5):615-6. No abstract available. PMID 4826961
- [Derived] Vain NE, Satragno DS, Gordillo JE, Fernandez AL, Carrolli G, Romero NP, Prudent LM. Postpartum use of oxytocin and volume of placental transfusion: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2020 Jan;105(1):14-17. doi: 10.1136/archdischild-2018-316649. Epub 2019 May 9. PMID 31072967
- See also: WHO recommendations — http://apps.who.int/rhl/evidence_summaries/beneficial/es/index.html